CLINICAL TRIAL: NCT00444873
Title: A Phase III, Multicentre, Open Label, Comparative, Dose-interval Titration Study Evaluating the Efficacy and Safety of Six Repeated Deep Subcutaneous Administrations of Lanreotide Autogel 120mg, in Acromegalic Patients Previously Treated With Octreotide LAR
Brief Title: Effect of 120mg Somatuline Autogel at Different Dose Intervals (28, 42 or 56 Days) in Patients With Acromegaly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-94-52030-163; 2004-001435-33 (EudraCT Number)
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Acromegaly
Keywords: Inappropriate Growth Hormone Secretion Syndrome (Acromegaly)
MeSH Terms: conditions — Acromegaly | interventions — lanreotide; Duration of Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 28 day dose interval (Experimental)
  Interventions: Drug: lanreotide (Autogel formulation), duration of treatment 24-56 weeks, depending on dose interval
- 42 day dose interval (Experimental)
  Interventions: Drug: lanreotide (Autogel formulation), duration of treatment 24-56 weeks, depending on dose interval
- 56 day dose interval (Experimental)
  Interventions: Drug: lanreotide (Autogel formulation), duration of treatment 24-56 weeks, depending on dose interval

INTERVENTIONS:
Drug: lanreotide (Autogel formulation), duration of treatment 24-56 weeks, depending on dose interval — Six deep subcutaneous injections of Lanreotide Autogel, 24-56 week intervals.

SUMMARY:
A multicentre, prospective, open label study of acromegalic patients evaluating the efficacy and safety of different dose-intervals of Lanreotide Autogel 120mg according to international standards and compared to previous treatment with Octreotide LAR 10, 20 or 30 mg.

DETAILED DESCRIPTION:
Six repeated applications of Lanreotide Autogel 120mg administered every 28, 42 or 56 days. For the first three injections, the interval depends on the Octreotide LAR dosage administered previously. The dose interval is titrated after injection 3 depending on the efficacy of the therapy with Lanreotide Autogel

ELIGIBILITY:
Inclusion Criteria:

* The patient must give written (personally signed and dated) informed consent before completing any study-related procedure.
* The patient must have a documented diagnosis of active acromegaly and be adequately treated with a stable dose (10, 20 or 30 mg) of Octreotide LAR for at least 6 months immediately prior to study entry. A documented diagnosis of active acromegaly is defined as IGF-1 more than 30% higher than two Standard Deviations ( +2 SD) above the normal age and sex adjusted value (see Appendix 6) or GH level after OGTT (Oral Glucose Tolerance Test) > 2ng/mL while not under drug treatment for acromegaly. For patients having undergone surgery or radiotherapy, this diagnosis must have been performed after the most recent surgical or radiation treatment

Exclusion Criteria:

* The patient has had pituitary surgery (adenomectomy) within 6 months prior to study entry
* The patient has received stereotactic (LINAC, Gamma Knife) radiotherapy for acromegaly within three years or conventional radiotherapy for acromegaly within five years prior to study entry

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Mean Insulin like Growth Factor 1 (IGF-1) and Growth Hormone (GH) levels at the beginning and end of the study and as proportion of patients conforming to internationally accepted levels. | 1 dose interval after the last administration of Lanreotide Autogel 120mg

SECONDARY OUTCOMES:
Dose interval, 28, 42 or 56 days for repeated injections of Lanreotide Autogel 120mg which are effective in reducing IGF-1 and GH levels to internationally accepted levels. | Last three injections of Lanreotiude Autogel 120mg
Dose interval, 28, 42 or 56 days for repeated injections of Lanreotide Autogel 120mg, which shows comparable efficacy to the previous treatment with Octreotide LAR 10, 20 or 30 mg in controlling IGF-1 and GH levels | Interval between doses after titration in part 2 of treatment (injections 3-6)
Patient symptoms and quality of life on Lanreotide Autogel and comparison to previous Octreotide LAR treatment. | 1 dose interval after the last administration of Lanreotide Autogel 120mg

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Klinikum Innenstadt, Munich, Germany

REFERENCES:
- [Result] Schopohl J, Strasburger CJ, Caird D, Badenhoop K, Beuschlein F, Droste M, Plockinger U, Petersenn S; German Lanreotide Study Group. Efficacy and acceptability of lanreotide Autogel(R) 120 mg at different dose intervals in patients with acromegaly previously treated with octreotide LAR. Exp Clin Endocrinol Diabetes. 2011 Mar;119(3):156-62. doi: 10.1055/s-0030-1267244. Epub 2010 Nov 17. PMID 21086246